CLINICAL TRIAL: NCT03288298
Title: Therapeutic Effect Of Luteolin Natural Extract Versus Its Nanoparticles On Tongue Squamous Cell Carcinoma Cell Line: In Vitro Study
Brief Title: Therapeutic Effect Of Luteolin Natural Extract Versus Its Nanoparticles On Tongue Squamous Cell Carcinoma Cell Line
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Safaa Elbaz, Assistant Lecturer, Oral and Maxillofacial Pathology, BUE, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEBD-CU-2017-09-23
Record Dates: First submitted 2017-09-12; First posted 2017-09-20 (Actual); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Tongue Neoplasms; Carcinoma
Keywords: TSCC; OSCC; luteolin; nanoluteolin; nanotechnology; oral cancer; apoptosis; PCR; MTT; ELISA reader
MeSH Terms: conditions — Tongue Neoplasms; Carcinoma; Mouth Neoplasms | interventions — Luteolin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- luteolin (Experimental): a natural extract derived flavinoids
  Interventions: Drug: luteolin
- nano-luteolin (Active Comparator): nano-particles derived from a natural extract luteolin
  Interventions: Drug: nano-luteolin

INTERVENTIONS:
Drug: luteolin — flavonoid natural extract
  Other Names: 3',4',5,7-tetrahydroxyflavone
  Arms: luteolin
Drug: nano-luteolin — nanoparticles of luteolin
  Other Names: nanoluteolin
  Arms: nano-luteolin

SUMMARY:
In vitro study to examine whether luteolin and nano-luteolin exert an inhibitory effect on tongue squamous cell carcinoma cell line by inducing apoptosis, and to assess if nano-luteolin has more efficient apoptotic activity than luteolin on tongue squamous cell carcinoma cell line.

DETAILED DESCRIPTION:
This study is conducted to examine whether luteolin and nano-luteolin exert an inhibitory effect on tongue squamous cell carcinoma cell line by inducing apoptosis, and to assess if nano-luteolin has more efficient apoptotic activity than luteolin on tongue squamous cell carcinoma cell line. The primary outcome is apoptosis, while the secondary outcome is cell viability.

ELIGIBILITY:
Inclusion Criteria:

* Squamous cell carcinoma cell lines (OSCC, TSCC and HNSCC).
* Luteolin 5,7,3',4'-tetrahydroxy-flavone (MeSH term).
* Application of luteolin as a chemotherapeutic drug.

Exclusion Criteria:

* Any cancer cell line other than OSCC, TSCC and HNSCC cell lines.
* Luteolin glycosides.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2018-09-01 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
gene expression of Caspase 3 to detect apoptosis | 6 hours
  fold-changes

SECONDARY OUTCOMES:
cell viability | 6 hours
  micromolar

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elkhadem, PhD, Study Chair — Center for Evidence Based Dentistry

REFERENCES:
- [Background] Ding S, Hu A, Hu Y, Ma J, Weng P, Dai J. Anti-hepatoma cells function of luteolin through inducing apoptosis and cell cycle arrest. Tumour Biol. 2014 Apr;35(4):3053-60. doi: 10.1007/s13277-013-1396-5. Epub 2013 Nov 28. PMID 24287949

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-18): https://cdn.clinicaltrials.gov/large-docs/98/NCT03288298/Prot_SAP_000.pdf